CLINICAL TRIAL: NCT06096402
Title: Selective Anterior Gastropexy as a Surgical Treatment Option for Paraesophageal Hernia
Brief Title: Gastropexy as a Treatment Option for Paraesophageal Hernia
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Collaborators: Hvidovre University Hospital (Other); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Kim Erlend Mortensen, MD, PhD, University Hospital of North Norway
Other Study IDs: 625668 (REK)
Record Dates: First submitted 2023-09-19; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Paraesophageal Hernia
Keywords: paraesophageal hernia; gastropexy; fundoplication
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anterior gastropexy, no fundoplication: patients with indication of operative management of a paraesophageal hernia
  Interventions: Procedure: no intervention, but surgical practice as usual is continued. Its a pragmatic study
- anterior gastropexy and fundoplication: patients with indication of operative management of a paraesophageal hernia
  Interventions: Procedure: no intervention, but surgical practice as usual is continued. Its a pragmatic study

INTERVENTIONS:
Procedure: no intervention, but surgical practice as usual is continued. Its a pragmatic study — no intervention

SUMMARY:
The present proposal aims to asses which is the optimal treatment strategy in a clinical study in patients with paraoesophageal hernia (PEH), a condition often found in elderly, fragile patients The investigator want to study the optimal approach to a paraoesophageal hernia (PEH) repair. The incidence of PEH increases with age and the older patient typically has additional co-morbidities, reduced physiological fitness, and frailty which makes surgery challenging regarding increased morbidity and mortality. Thus, the decision to offer surgery can be challenging in this cohort of patients. The need of an anti-reflux procedure as part of the repair is one of the main subjects for discussion worldwide. To date no consensus exists and many surgical centres do a routine anti-reflux procedure as part of their standard operation for PEH. But is this procedure redundant? Can the patients be managed with a less complicated procedure; an anterior gastropexy with comparable outcome?

DETAILED DESCRIPTION:
A hiatal hernia is a widening of the diaphragmatic hiatus causing herniation of the stomach into the thoracic cavity. It develops because of an insufficiency of the hiatus. The paraesophageal hernias (PEH) are classified as grade II-IV hiatal hernia with at least 50 % of the stomach misplaced in the thoracic cavity.

A paraesophageal hernia (PEH) is a potentially dangerous condition. One see in varied degree, the stomach and other organs being misplaced above diaphragm, in the thoracic cavity. Symptoms such as dysphagia, vomitus, weight loss, pain, short breath and emergent situations where abdominal organs are strangulated with risk of tissue death in thorax defines whether a patient should be offered operation and how fast it should be performed.

The operative management of PEH has become a laparoscopic procedure within the last 20-30 years with a concomitant significant decrease in morbidity and length of hospital stay. It is managed by different subspecialized surgeons, all of them having different perspectives and approaches to this condition. Surgery in this area is potentially high-risk operations with risk of perforation of oesophagus, injury to lungs, aorta, pericardia, spleen and stomach. Without operation symptomatic patients with PEH are at risk of developing an acute surgical condition with organ perforation with high per-and postoperative mortality.

Contemporary surgical technique is divided into three crucial steps; 1) removal of the hernia sac, 2) hiatoplasty with or without mesh and 3) an anti-reflux procedure and/or gastropexy. Each step is managed differently among surgeons/centres worldwide with varying evidence. Many surgeons add an anti-reflux procedure to the surgical management of PEH, to protect against postoperative acid reflux. The argument is that an anti-reflux procedure lowers postoperative reflux and recurrence of the paraesophageal hernia, but this is without clear evidence. As an addition or an alternative in step three of the PEH procedure, some centres do an anterior gastropexy to anchor the stomach in the abdominal cavity. It is a simple technique compared with an anti-reflux procedure with possibly equal satisfactory long-term outcomes but less postoperative complications. However, evidence is sparse and larger studies on this technique are highly warranted.

The aim is to study the need of a fundoplication as part of the procedure for PEH regarding symptom control and quality of life. For this reason, The investigator want to set up a prospective two-armed multicenter study in collaboration with St. Olav's Hospital, Trondheim and Gastroenheden, Hvidovre, Denmark. The reason for this collaboration is 1) to enlarge the group of investigation, as PEH is a rare condition, 2) to compare current practice (fundoplication/no fundoplication) among the included institutions. .

ELIGIBILITY:
Inclusion Criteria:

- Both emergent and elective repair of the paraoesophageal hernia

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with a paraesophageal hernia with indication of operation
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
peri- and postoperative complications | 30 days after operation
  according to clavien-dindo score
Gastro-esophageal reflux disease-Health related quality of life, GERD-HRQL | Before surgery and 3,6 and 12 months after surgery
  The GERD-HRQL questionnaire evaluates heartburn, dysphagia and regurgitation on a scale from zero (no symptoms) to five (severe symptoms) in 15 questions. Maximum score ranges from zero to 75 points
Short From questionnaire (SF-36) Health related quality of life | before surgery and 3, 6 and 12 months after surgery
  SF-36 is a well-established questionnaire consisting of 36 health related questions. Scale is from 0-100 for each section (8 sections) A high score corresponds to a better health status

SECONDARY OUTCOMES:
Total number of patients with radiological recurrence after one year | one year after surgery
  esophagus x-ray/barium swallow one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kim Erlend Mortensen, MD, PhD, Study Director — University of North Norway
Locations (3):
- Hvidovre Hospital, Copenhagen, Denmark
- Norway (2):
  - University Hospital of North Norway, Harstad
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided